CLINICAL TRIAL: NCT04419415
Title: Breakfast for Female Adolescent - NewStart
Acronym: NewStart
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: covid-19 lock down
Sponsor: University of Aarhus (Other)
Collaborators: The Danish Dairy Research Foundation, Denmark (Other)
Responsible Party: Principal Investigator, Mette Hansen, Associate professor, University of Aarhus
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: ProteinLab_P9_NyStart
Record Dates: First submitted 2020-03-13; First posted 2020-06-05 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Overweight Adolescents; Metabolic Disease
MeSH Terms: conditions — Metabolic Diseases | interventions — Breakfast; Exercise

STUDY DESIGN:
Intervention Model Description: 2x2 design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Skipping breakfast and maintain habitual physical activity (Experimental): Subject will skip breakfast and maintain habitual physical activity.
  Interventions: Other: Skipping breakfast
- High protein breakfast and maintain habitual physical activity (Experimental): Subject will consume a high protein dairy breakfast (300 g high protein yoghurt (skyr)) and maintain habitual physical activity.
  Interventions: Dietary Supplement: Breakfast with high protein dairy; Other: Skipping breakfast
- Skipping breakfast and exercising three times per week (Experimental): Subject will skip breakfast and participate in organized exercise-training three times per week (and maintain habitual physical activity)
  Interventions: Other: Exercise training
- High protein breakfast and exercising three times per week (Experimental): Subject will consume a high protein dairy breakfast (300 g high protein yoghurt (skyr)) and and participate in organized exercise-training three times per week (and maintain habitual physical activity)
  Interventions: Dietary Supplement: Breakfast with high protein dairy; Other: Exercise training

INTERVENTIONS:
Dietary Supplement: Breakfast with high protein dairy — High protein yoghurt containing approx. 10 g protein per 100 g. Participants will be asked to consume 300 g (=3 dl) for breakfast.
  Arms: High protein breakfast and exercising three times per week; High protein breakfast and maintain habitual physical activity
Other: Exercise training — Participants will be asked to participate in organized exercise training 3 times per week.
  Arms: High protein breakfast and exercising three times per week; Skipping breakfast and exercising three times per week
Other: Skipping breakfast — Participants will be asked to skip breakfast.
  Arms: High protein breakfast and maintain habitual physical activity; Skipping breakfast and maintain habitual physical activity

SUMMARY:
Investigators will test the long-term health effects of eating a dairy-based protein-rich breakfast and/or performing regular physical training for 12 weeks in 100 previous 'breakfast skipping' young overweight women (2 x 2 factorial design). Measurements of body composition, physical fitness, metabolic health parameters, faeces (microbiota activity and composition), satiety and daily energy intake will be collected.

DETAILED DESCRIPTION:
The study is a 2×2-factorial randomized controlled trial with 4 study arms. The subjects will be randomly allocated to skip breakfast or eat high-protein yoghurt products (300g/day) and to either exercise 3x per week or maintain habitual physical activity for 12 weeks. Measurements and biological sampling will be performed at baseline and at the end of the intervention period.

The primary outcome will be fat mass and fat free mass. The investigators will also measure effects on weigth, waiste, health-related blood paramenters, muscle function, metabolites in urine and blood, and gut microflora and pH.

ELIGIBILITY:
Inclusion Criteria:

* BMI >25
* exercising < 1 h per week.

Exclusion Criteria:

* smoking
* illness and use of medication affecting the study outcomes
* allergy towards milk and yoghurt
* weightloss/gain >5kg the last 6 months
* dieting
* eating disorder
* pregnancy
* breast feeding
* unable to speak and understand danish

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Body composition (DXA scan) 1 | 12 weeks
  Fat mass in grams
Body composition (DXA scan) 2 | 12 weeks
  Fat free mass in grams

SECONDARY OUTCOMES:
HbA1c | 12 weeks
  Blood sample measurement of HbA1c
LDL | 12 weeks
  Blood sample measurement of LDL
HDL | 12 weeks
  Blood sample measurement of HDL
Health related blood parameter 1 | 12 weeks
  blood sample measurement of fasting glucose
Health related blood parameter 2 | 12 weeks
  Blood sample measurement of fasting insulin
Health related parameter | 12 weeks
  Oral glucose tolerance test measured as the area under the curve
Fitness | 12 weeks
  Aastrand bike test
Muscle strength | 12 weeks
  grib strength (kg)
maximal jump height | 12 weeks
  maximal jump height (cm)
weight | 12 weeks
  Body weight (kg)
Height | 12 weeks
  Body hight (m)
BMI | 12 weeks
  weight measurement in kg, height in meters
Food log | 12 weeks
  4-day food log (energy in KJ)
Gut microflora | 12 weeks
  by bacterial determination of faeces
Feaces pH | 12 weeks
  by pH determination of faeces
Urine metabolites | 12 weeks
  by metabolomics
Blood metabolites | 12 weeks
  by metabolomics

CONTACTS AND LOCATIONS:
Overall Officials: Mette Hansen, PhD, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Department for Public Health, Section for Sport Science, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No